CLINICAL TRIAL: NCT06129409
Title: A Randomized, Double -Blind (Sponsor-Open), Placebo-Controlled Study to Assess the Effect of NT-0796 on Inflammation in Obese Participants at Risk of Cardiovascular Disease
Brief Title: Effects of NT-0796 in Obese Participants at Risk of Cardiovascular Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NodThera Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NT-0796-P003
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Drug vs Placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT-0796 (Experimental): BID
  Interventions: Drug: NT-0796
- Placebo (Placebo Comparator): BID
  Interventions: Drug: NT-0796

INTERVENTIONS:
Drug: NT-0796 — Orally administered capsules

SUMMARY:
This trial is a Randomized, Double-Blind (Sponsor-Open), Placebo-Controlled Study to Assess the Effect of NT-0796 on Inflammation in Obese Participants at Risk of Cardiovascular Disease.

Participants will be admitted to an in-patient Clinical Research Unit on Day -1 and will be discharged on Day 30. The trial will include a 7-day out-patient safety follow-up period following the last dose of study treatment.

For the first approximately 20 participants effect of food will be evaluated on the Pharmacokinetics of NT-0796. MRI's will be conducted in a subset of participants.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effects of NT-0796 on inflammation in obese participants at risk of cardiovascular disease, evaluate the effects of NT-0796 on body weight and composition, to see how safe NT-0796 is, and how well it is tolerated and to measure the blood levels of NT-0796, with and without food.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older.
2. Body mass index (BMI) ≥30 and ≤40 kg/m2 at screening.
3. Presence of 1 or more of the following risk factors for atherosclerotic cardiovascular disease:

   * History of controlled hypertension
   * History of hypercholesterolemia
   * History of high-density lipoprotein levels
   * Controlled Type 1 or Type 2 Diabetes mellitus

Exclusion Criteria:

1. History of stroke with residual neurological deficit within 2 years or transient ischemic attack within 6 months
2. History of acute coronary syndrome (ACS)
3. Stable angina.
4. Diagnosis of congestive heart failure
5. Evidence of past or current infection with Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in hsCRP levels | Baseline to Day 28
  Evaluate the effects of NT-0796 on inflammation.

SECONDARY OUTCOMES:
Change in Body weight (kg) | Change from baseline to Day 28
Body composition | Change from baseline to Day 28
  Absolute Fat mass, % Body Fat and Visceral Fat (L)

OTHER OUTCOMES:
Clinical laboratory values | Change from baseline to Day 28
  Haematology and Clinical Chemistry
Vital signs | Change from baseline to Day 28
  Body temperature, heart rate and systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Investigative Site, Miami, Florida
  - Investigative Site, Austin, Texas